CLINICAL TRIAL: NCT05899244
Title: Determining the Most Efficient Techniques of Gain of Range of Motion in Function of the Type of Limitation in Asymptomatic Subjects.
Brief Title: Influence of Muscle Stretching and Neural Mobilizations on Lower Limbs Range of Motion in Asymptomatic Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Pesesse Pierre, Physiopherapist PHD student, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ULiège Pesesse Pierre 02
Record Dates: First submitted 2023-04-05; First posted 2023-06-12 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Asymptomatic Condition
Keywords: Straight leg raising test; Knee extension angle; Neural mobilization; Muscle Stretching; Asympotmatic subject
MeSH Terms: conditions — Asymptomatic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor is blind to participant group allocation. After the first evaluation participant are conduct in another room where a second investigator allocate them to a subgroup and give them instructions concerning the intervention. After a month the re-avaluation takes place and patient are told to keep secret their affiliation group until the end of the re-evaluation in order to keep the outcomes assessor blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Muscle limitation subgroup receiving muscle stretching exercice (Experimental): This subgroup of participants will have to perform 2 muscle stretching exercices every day during a month and to report the frequency of realisation on a smartphone or a web application.
  Interventions: Other: muscle streching exercice
- Muscle limitation subgroup receiving a slider exercice (Experimental): This subgroup of participants will have to perform two series of ten repetitions of a slider exercice every day during a month and to report the frequency of realisation on a smartphone or a web application.
  Interventions: Other: Slider
- Muscle limitation subgroup receiving a tensioner exercice (Experimental): This subgroup of participants will have to perform two series of ten repetitions of a tensioner exercice every day during a month and to report the frequency of realisation on a smartphone or a web application.
  Interventions: Other: Tensioner
- Neural limitation subgroup receiving a muscle stretching exercice (Experimental): This subgroup of participants will have to perform 2 muscle stretching exercices every day during a month and to report the frequency of realisation on a smartphone or a web application.
  Interventions: Other: muscle streching exercice
- Neural limitation subgroup receiving a slider exercice (Experimental): This subgroup of participants will have to perform two series of ten repetitions of a slider exercice every day during a month and to report the frequency of realisation on a smartphone or a web application.
  Interventions: Other: Slider
- Neural limitation subgroup receiving a tensioner exercice (Experimental): This subgroup of participants will have to perform two series of ten repetitions of a tensioner exercice every day during a month and to report the frequency of realisation on a smartphone or a web application.
  Interventions: Other: Tensioner
- Neural limitation Control subgroup (No Intervention): Participants in this subgroup will not receive an intervention.
- Muscle limitation Control subgroup (No Intervention): Participants in this subgroup will not receive an intervention.

INTERVENTIONS:
Other: muscle streching exercice — For this exercice the participant will have to place the foot of the stretched leg on a step while maintaining his knee in extension.
  From this starting position the patient will have to do a pelvic anterior tilt while keeping is back straight and his gaze horizontal until the movement induce a feeling of stretching in the posterior part of the thigh.
  Arms: Muscle limitation subgroup receiving muscle stretching exercice; Neural limitation subgroup receiving a muscle stretching exercice
Other: Slider — In order to define the starting position for a slider, the participant will be positioned in lateral decubitus with the knee extended and will perform a hip flexion until a sensation of pain or stretching feeling appears on the posterior part of the thigh or of the knee. If the hip flexion does not induce a stretching sensation or pain, a dorsal ankle flexion is added. Once this position is defined the patient slightly reduces the amount of hip flexion until the stretching/pain sensation disappears.
  From this starting position, to perform the slider: the subject performs a hip flexion movement and simultaneously a cervical extension movement, this corresponds to the outward movement. For the return movement the patient performs a hip extension and at the same time a cervical flexion. The slider technique must be pain free.
  Other Names: neural sliding mobilization
  Arms: Muscle limitation subgroup receiving a slider exercice; Neural limitation subgroup receiving a slider exercice
Other: Tensioner — The participant will be positioned in lateral decubitus with the knee extended and the hip, the cervical, thoracic and lumbar spine placed in neutral position.
  For the outward movement, the participant will perform a hip flexion associated with a simultaneous movement of cervical extension until a sensation of pain or a stretching feeling appears on the posterior part of the thigh or of the knee.If this combined movements do not induce a stretching sensation or pain, a dorsal flexion of the ankle is added.
  For the return movement, the participant will realize a hip extension simultaneously associated to a movement of extension of the cervical spine. If the dorsal flexion of the ankle was used during the outward movement, a movement plantar flexion of the ankle must be used in association to the movement of hip extension.
  Other Names: neural tensioning mobilization
  Arms: Muscle limitation subgroup receiving a tensioner exercice; Neural limitation subgroup receiving a tensioner exercice

SUMMARY:
First, this study aims to use the straight leg raising test (SLR) and the knee angle extension test (KEA) test associated to a structural differentiation to determine the limitation of the lower limb (muscular or nervous) in asymptomatic subjects.

Second, this study will try to determine the most efficient exercice to increase range of motion of the lower limb in function of subjects limitation type (muscular, nervous,) using neural mobilization (sliders or tensioners) and muscle stretching.

Two groups will be constituted for each test (SLR and KEA) based on the limitation defined during the test:

Group 1: Muscle limitation Group 2: Neural limitation

Each group will be subdivided in four subgroups depending on the intervention participants will receive:

* subgroup 1: Muscle stretching group
* subgroup 2: Neural tensioner group
* subgroup 3: Neural slider group
* subgroup 4: Control group

Participants from groups 1,2 and 3 will be asked to do an exercice every day during 31 days, independently of their subgroup allocation.

Participants from group 1 will perform a muscle stretching technique during 20 second twice a day.

Participants from group 2 will do 10 repetitions of tensioner twice a day. Participants from group 3 will do 10 repetitions of a slider twice a day.

Subgroup comparisons of the evolution of the range of motion during SLR and KEA before and after the month of exercice will determine which technique is the most efficient for a specific type of limitation.

DETAILED DESCRIPTION:
Objectives:

First, this study aims to use the straight leg raising test (SLR) and the knee angle extension test (KEA) test associated to a structural differentiation to determine the limitation of the lower limb (muscular or nervous) in asymptomatic subjects.

Second, this study will try to determine the most efficient exercice to increase range of motion of the lower limb in function of subjects limitation type (muscular, nervous,) using neural mobilization (sliders or tensioners) and muscle stretching.

Procedures:

All the participants will attend two assessment sessions i.e., at baseline and after 31 days, expect for participants allocate in the control group, who will be also tested 48 to 72 hours after the first evaluation in order to determine the test/retest reliability of the structural differentiation.

Baseline session:

During the baseline session, demographics data will be collected (age, gender, height and weight) and a check for exclusions criteria will be conducted. The identification of the dominant lower limb will then be performed by asking participants to shoot on a ball

The Identification of the limitation

The leg to be tested will be the dominant one in half of the population while the other half will have the non-dominant leg tested. In order to standardize the assessments, participants will be placed supine with the cervical spine in neutral position and with the upper part of head at the edge of the examination table (Table with a moveable head set) with both hands placed under the lumbar spine. Furthermore, a belt will be place to fix the pelvis to the examination table at the level of the anterior superior iliac spine.

The SLR and the KEA tests will then be performed. For standardization purposes, the same sequence of testing will be used at each session for the same participant (first SLR and second KEA or conversely), but sequences of tests will be used alternatively between participants to avoid methodological bias. Participants will be asked to say "stop" when a discomfort appears at the posterior part of the tight, the calf, the knee, the buttock or in the foot.

For the SLR, the investigator will induce a hip flexion movement, while maintaining the knee in extension, with one hand placed on the distal anterior part of the tight and with the other hand located on the posterior distal part of the leg (9).

For the KEA a labrique inclinometer will be placed on the anterior part of the tight allowing the investigator to control that a 90° of hip flexion is maintained, while he will passively induce a knee extension.

A second investigator will evaluate the hip and knee range of motion during the SLR and KEA respectively, with an electronical inclinometer using the more proximal part of the tibial tuberosity as a marker for the device placement.

While maintaining the ipsilateral SLR or KEA, a structural differentiation (SD) will be used to identify the structure related to patient discomfort. In order to do the SD, 2 stages will be conducted: first a third investigator will passively induce a flexion of the thoracic spine using the movable cranial part of the table and will manually move the cervical spine in flexion. The participant will then be invited to define if the discomfort in the limb tested is modified using the following predefined descriptors: increase, decrease, not changed, different location of the symptoms or a combination of these. In the second stage, the third investigator will induce a passive extension of the thoracic and cervical spine and participants will be asked to report any potential changes of the lower limbs discomfort using the same descriptors as mentioned previously.

Interpretation of the tests and group allocation:

If both stages of the SD did not change the lower limb discomfort, a "muscle limitation" will be suspected. Nervous structures will be suspected to be the limiting factor, if the discomfort was increased during the flexion part of the SD and decreased during the extension part.

Thereby, participants will be divided in two groups: the "Nerve group"will included the participants in whom nervous structures were suspected to be the limiting factor after SD ; the "Muscle group" will include participant for whom a "muscle limitation" was suspected.

Exercise allocation will be done by another investigator in a separate room. In each groups ("Nerve" or "Muscle"), participants will be randomized in one of the four following subrgroups:

* subgroup 1: Muscle stretching group
* subgroup 2: Neural tensioner group
* subgroup 3: Neural slider group
* subgroup 4: Control group

Participants from groups 1,2 and 3 will be asked to do an exercice every day during 31 days, independently of their subgroup allocation.

Participants from group 1 will perform a muscle stretching technique during 20 second twice a day.

Participants from group 2 will do 10 repetitions of tensioner twice a day. Participants from group 3 will do 10 repetitions of a slider twice a day.

Subgroup comparisons of the evolution of the range of motion during SLR and KEA before and after the month of exercice will determine which technique is the most efficient for a specific type of limitation.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Asymptomatic subject

Exclusion Criteria:

* Mutiple Sclerosis
* diabetis
* Neuropathy
* Stroke
* Lumbar pain during the last 6 month
* Lumbosacral radicular pain
* Meningitis
* Sequelae of hamstring, gluteal or sural triceps tear
* Sequelae of Achilles tendon section
* Guillain-Barré Syndrom
* hip and Knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

PRIMARY OUTCOMES:
Change of the limitation type during the Knee extension angle test (KEA) after 31 days | After 31 days
  This outcome will be definfed as a muscle limitation or as a nerve limitation using the structural differentiation.
Change of Knee extension range of motion during KEA after 31 days | After 31 days
  This outcome corresponds to the angle of Knee extension mesured during the KEA which induced a discomfort or an unpleasant feeling at the posterior part of the buttock, the thigh, the leg or in the foot reported by the participant.
  An electronical inclinometer will be used for the measurement of this angle, placed on the tibial bone using the anterior tibial tuberosity as a reference point.
Change of limitation type of during the Straight leg raising test (SLR) after 31 days | After 31 days
  This outcome will be definfed as a muscle limitation or as a nerve limitation using the structural differentiation.
Change of Hip flexion range of motion during the Straight leg raising test after 31 days | After 31 days
  This outcome corresponds to angle of hip flexion measured during SLR test which induced a discomfort or an unpleasant feeling at the posterior part of the buttock, the thigh, the leg or in the foot reported by the participant.
  An electronical inclinometer will be used for the measurement of this angle, placed on the tibial bone using the anterior tibial tuberosity as a reference point.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Pesesse, master, Principal Investigator — University of Liege
Locations (1):
- UNiversity of liege, Liège, Liege, Belgium

IPD SHARING:
Plan to Share IPD: No